CLINICAL TRIAL: NCT01767948
Title: An Open-Label, Multicenter, Pharmacokinetic Study of PCI-32765 in Subjects With Varying Degrees of Hepatic Impairment
Brief Title: A Study to Evaluate the Pharmacokinetics of PCI-32765 in Participants With Varying Degrees of Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR100944; PCI-32765CLL1006 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2013-01-09; First posted 2013-01-15 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Hepatic Impairment
Keywords: Hepatic Impairment; PCI 32765; Metabolite PCI-45227; Pharmacokinetics
MeSH Terms: interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Patients with mild hepatic function (Experimental): Patients will receive PCI-32765 140 mg, orally, as a single dose, on Day 1.
  Interventions: Drug: PCI-32765
- Patients with moderate hepatic function (Experimental): Patients will receive PCI-32765 140 mg, orally, as a single dose, on Day 1.
  Interventions: Drug: PCI-32765
- Patients with severe hepatic function (Experimental): Patients will receive PCI-32765 140 mg, orally, as a single dose, on Day 1.
  Interventions: Drug: PCI-32765
- Patients with normal hepatic function (Experimental): Patients will receive PCI-32765 140 mg, orally, as a single dose, on Day 1.
  Interventions: Drug: PCI-32765

INTERVENTIONS:
Drug: PCI-32765 — PCI-32765 140 mg will be administered as a single dose, orally, on Day 1.

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (how the drug concentrations change over time) of PCI 32765 in participants with mild, moderate, or severe hepatic impairment.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), single-dose, multi-center (study conducted at multiple sites), non-randomized study to access the pharmacokinetics of PCI-32765 in participants who either have mild, moderate, or severe hepatic impairment or qualify for the control group (normal liver function). The study mainly consists of 3 phases: screening phase (within 21 days prior to the first dose of study medication), treatment phase, and a follow up phase (10 to 12 days after the last dose of study medication). In the treatment phase, participants will receive single oral dose of PCI-32765 on Day 1. Liver impairment will be classified according to the Child-Pugh Classification of Severity of Liver Disease, as: normal, mild, moderate, and severe. Total 30 participants (24 with hepatic impairment [6 mild, 9 moderate and 9 severe] at baseline and 6 in the control group according to Child-Pugh criteria) will be enrolled. Participants in the control group will be enrolled after the participants with mild or moderate hepatic impairment have completed the study. Safety evaluations for adverse events, clinical laboratory tests, electrocardiogram, vital signs, and physical examination will be monitored throughout the study. The total duration of study for each participant will be approximately for 29 to 33 days.

ELIGIBILITY:
Inclusion Criteria:

* Stable hepatic function as confirmed by the serum bilirubin and transaminase levels measured during screening and those measured within 48 hours prior to PCI-32765 administration
* Must be hepatically impaired as defined by the Child-Pugh classification of severity of liver disease
* Control group must have good health with normal liver function
* Participants with controlled hypertension and those with problems directly associated with the primary diagnosis of hepatic impairment
* Concomitant medications to treat underlying disease states or medical conditions related to hepatic impairment are allowed
* Agrees to protocol-defined use of effective contraception

Exclusion Criteria:

* Clinically significant renal laboratory findings including serum creatinine more than 1.5 x the upper limit of normal (ULN) and/or calculated creatinine clearance of less than 60 ml per minute per 1.73 square meter
* Clinically significant abnormal laboratory tests, physical examination, vital signs or electrocardiogram at screening or at admission to the study center
* Antiviral therapy for active hepatitis infection at time of screening
* Use of any anti-coagulation therapy including vitamin K antagonists, low molecular weight heparin, or other anticoagulants

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration of PCI-32765 | Predose, 30 minutes, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 16 hours, 24 hours, 36 hours, 48 hours, 72 hours, and 96 hours
Area under the plasma concentration of PCI-32765 | Predose, 30 minutes, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 16 hours, 24 hours, 36 hours, 48 hours, 72 hours, and 96 hours

SECONDARY OUTCOMES:
Number of participants with adverse events | up to Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical trial, Study Director — Janssen Research & Development, LLC
Locations (4):
- United States (4):
  - Costa Mesa, California
  - Orlando, Florida
  - Knoxville, Tennessee
  - San Antonio, Texas

REFERENCES:
- [Derived] de Jong J, Skee D, Hellemans P, Jiao J, de Vries R, Swerts D, Lawitz E, Marbury T, Smith W, Sukbuntherng J, Mannaert E. Single-dose pharmacokinetics of ibrutinib in subjects with varying degrees of hepatic impairment<sup/> Leuk Lymphoma. 2017 Jan;58(1):185-194. doi: 10.1080/10428194.2016.1189548. Epub 2016 Jun 7. PMID 27267254
- See also: An Open-Label, Multicenter, Pharmacokinetic Study of PCI-32765 in Subjects with Varying Degrees of Hepatic Impairment(18343). — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=3612&filename=CR100944_CSR.pdf